CLINICAL TRIAL: NCT01864707
Title: Randomized Controlled Trial on the Efficacy of Acupuncture and the Efficacy of Mindfulness-Based Stress Reduction (MBSR) in Patients With Multiple Sclerosis Suffering From Fatigue
Brief Title: Acupuncture or MBSR for Patients With Fatigue and MS
Acronym: MS-Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia M. Witt, Prof. Dr. med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS-Fatigue-13
Record Dates: First submitted 2013-04-02; First posted 2013-05-30 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Fatigue; Multiple Sclerosis
Keywords: multiple sclerosis, fatigue
MeSH Terms: conditions — Fatigue; Multiple Sclerosis | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- usual care + acupuncture (Experimental): standardized acupuncture treatment in addition to usual care
  Interventions: Other: Usual care + acupuncture
- usual care+mbsr (Experimental): mindfulness based stress reduction in addition to usual care not recruiting anymore
  Interventions: Other: usual care+mbsr
- usual care (Active Comparator): usual care without additional treatment
  Interventions: Other: usual care

INTERVENTIONS:
Other: Usual care + acupuncture — Patients of this group receive a standardized acupuncture treatment over 12 weeks in addition to usual care
  Arms: usual care + acupuncture
Other: usual care+mbsr — Patients of this group receive mindfulness based stress reduction in addition to usual care
  Arms: usual care+mbsr
Other: usual care — Patients in this group will follow the same treatment for fatigue they received at study entry
  Arms: usual care

SUMMARY:
The main aim of this trial is to evaluate whether additional acupuncture or mindfulness-based stress reduction is more efficacious than usual care only to reduce fatigue in patients with multiple sclerosis.

DETAILED DESCRIPTION:
In multiple sclerosis, fatigue is the most common clinical symptom, reported by up to 97% of patients. No successful evidence-based therapy exists so far. The main aim of this trial is to evaluate whether additional acupuncture or mindfulness-based stress reduction is more efficacious than usual care only to reduce fatigue in patients with multiple sclerosis. We want to include 141 patients with multiple sclerosis and fatigue. Participants will be randomised into three groups to compare 1) usual care, 2) usual care plus standardised acupuncture, and 3) usual care plus mindfulness-based stress reduction. Treatment duration will be 12 weeks. The primary outcome is the Fatigue Severity Scale (FSS) after 12 weeks, follow-up measurement will be performed after 26 weeks. Secondary outcomes include other fatigue specific parameters, other MS specific parameters, cost, and physiological, immunological and functional magnetic resonance imaging parameters.

ELIGIBILITY:
Inclusion Criteria:

* female or male
* 18 to 65 years of age
* able to give oral and signed written informed consent
* clinical diagnosis of multiple sclerosis
* fatigue in "multiple sclerosis" for at least 3 months
* other stable pre-study treatment with respect to target symptom fatigue for at least 3 months before inclusion
* stable immunomodulatory or immunosuppressive therapy or stable no such a therapy for at least the 3 months before inclusion
* fatigue score of ≥4 on the Fatigue Severity Scale at inclusion
* patient's mental and physical ability to participate in the trial
* willingness to be randomised, to attend visits, to complete questionnaires, and willingness to participate and fMRI measurements

Exclusion Criteria:

* fatigue because of a malignant disease
* acute relapse or cortisone therapy therapy in the last 30 days before inclusion
* EDSS (Extended disability status scale) > 6
* fatigue specific acupuncture in the last 12 months
* during the last 12 months performing of MBSR exercises learnt in the past
* change of immunomodulatory or immunosuppressive therapy during the 3 months before inclusion
* other new therapies are planned which could have a positive effect on fatigue (e.g. exercise, acupuncture, relaxation therapy)
* for female patients: pregnancy or anticipated pregnancy during the intervention period
* severe acute and or chronic disease which does not allow participation in the therapy
* other limitations which do not allow participation in the therapy
* alcohol or substance abuse
* parallel participation in another clinical trial
* BDI > 29
* contra indications for fMRI session (e.g. metal clips)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2013-04; Primary Completion 2015-06 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
fatigue severity scale | 12 weeks

SECONDARY OUTCOMES:
fatigue severity scale | 26 weeks
modified fatigue impact scale | baseline, 8 weeks, 26 weeks
therapy response rates | 12 weeks
expanded disability status scale | baseline, 12 weeks, 26 weeks
multipe sclerosis functional composite scale | baseline, 12 weeks, 26 weeks
beck depression inventory II | baseline, 12 weeks, 26 weeks
Body efficacy expectation | baseline, 12 weeks, 26 weeks
  Body-Efficacy Expectation (BEE) is a scale to measure the conviction that one's body is able to deal with health-threatening factors by itself. It is a six items' scale developed in the Institute of Social Medicine, Epidemiology and Health Economics and not published, yet.
SF-12 | baseline, 12 weeks, 26 weeks
HAQUAMS | baseline, 12 weeks, 26 weeks
Costs | baseline, 12 weeks, 26 weeks
  Data on Resource-consumption and associated costs are planned to be derived as patient-reported information using the patient questionnaires.
overall treatment effect | 12 weeks, 26 weeks
immune parameters | baseline, 12 weeks, 26 weeks
  PBMC and proliferationsassays, pro- and antiinflamatory cytokines, axonal damage marker such as neurofilaments and neurotrophic factors like BDNF
  possible influences on the immune system will be evaluated in an exploratory way.
number of serious adverse events | 12 weeks, 26 weeks
number of suspected adverse reactions | 12 weeks, 26 weeks

OTHER OUTCOMES:
fMRI | baseline, 12 weeks, 26 weeks
  e.g. functional connectivity in a subgroup of 20 subjects in each group
Dynamics of saccade parameters | baseline, 12 weeks, 26 weeks, and directly after one acupuncture session
  Eye movement analysis will be performed according established standards (Finke et al, J Neurol 2012)
Qualitative interviews regarding therapy | 26 weeks
  Part of the patients will be interviewed about the therapies.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia M Witt, MD, Principal Investigator — Institute for Social Medicine, Epidemiology and Health Economics, Charité - Universitätsmedizin Berlin; Friedemann Paul, MD, Principal Investigator — The NeuroCure Clinical Research Center, Charité - Universitätsmedizin Berlin
Locations (1):
- The NeuroCure Clinical Research Center, Charité - Universitätsmedizin Berlin, Berlin, State of Berlin, Germany